CLINICAL TRIAL: NCT05517109
Title: The Influence of Different Hemodynamic Parameters in First 24 Hours After Intravenous Thrombolysis on Acute Ischemic Stroke Outcomes: a Randomised Clinical Trial
Brief Title: Hemodynamic in Postreperfusion Period and Functional Recovery in Acute Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IVT-160
Record Dates: First submitted 2022-08-06; First posted 2022-08-26 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke; Intracranial Hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group. Standart care (No Intervention): Standart hemodynamic goals: systolic blood pressure 160-185 mmHg in first 24 hours after intravenous thrombolysis
- Systolic blood pressure ≤ 160 mmHg (Experimental): Lower hemodynamic goals: systolic blood pressure ≤ 160 mmHg in first 24 hours after intravenous thrombolysis
  Interventions: Other: Hemodynamic goal including lower goal of systolic blood pressure

INTERVENTIONS:
Other: Hemodynamic goal including lower goal of systolic blood pressure — Different hemodynamic goals in different study arms
  Arms: Systolic blood pressure ≤ 160 mmHg

SUMMARY:
The investigators are suggtesting that lower goals of systolic blood pressure after intravenous thrombolysis may reduce the risk of hemorrhagic complications and improve functional outcomes after acute ischemic stroke.

ELIGIBILITY:
Inclusion сriteria:

* ischemic stroke diagnosis
* performed intravenous thrombolysis (including "wake up stroke")
* systolic blood pressure >140 mmHg
* informed consent or council of physician agreement

Exclusion criteria:

* absence of informed consent or council of physician agreement
* pregnancy
* patients participainting in other clinical trial in the last 90 days
* any absolute contraindications to intravenous thrombolysis

Сompletion criteria:

* failure to achieve hemodynamic goal for 20 minutes before the start of intravenous thrombolysis
* failure to achieve hemodynamic goal for 60 minutes in first 24 hours after intravenous thrombolysis
* relative arterial hypotension (SBP <100 mmHg for 60 minutes in first 24 hours after intravenous thrombolysis)
* unfavorable effect development (e.g. seizures, angioedema)
* informed consent is retracted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90 day after intravenous thrombolysis
  Fucntional outcome (Modified Rankin Scale) will be assesed by telephone interview. Score from 0 to 6. Higher scores mean a worse outcome.
Mortality rate | At 90 day after intravenous thrombolysis
Rate of symptomatic intracranial hemorrhage | 24 hours after intravenous thrombolysis
  Symptomatic intracranial hemorrhage (sICH) according to SITS-MOST study description of sICH
Rate of symptomatic intracranial hemorrhage | 7 days after intravenous thrombolysis
  Symptomatic intracranial hemorrhage (sICH) according to SITS-MOST study description of sICH

SECONDARY OUTCOMES:
Change in National Institutes of Health Stroke Scale (NIHSS) | at 28 day after intravenous thrombolysis
  Score form 0 to 42. Higher score indicates worse outcome
Rate of all Intracranial hemorrhage | 24 hours after intravenous thrombolysis
  Intracranial hemorrhage will be classified according to Heidelberg bleeding classification
Rate of all Intracranial hemorrhage | 7 days after intravenous thrombolysis
  Intracranial hemorrhage will be classified according to Heidelberg bleeding classification
Lengths of stay in ICU | at 90 day after intravenous thrombolysis
Lengths of stay in hospital | at 90 day after intravenous thrombolysis
Rate of acute kidney injury | 28 day after intravenous thrombolysis or at discharge
  Acute kidney injury will be assesed according to RIFLE Classification

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kirov, PhD, Study Director — Northen state medical university; Alexey Avidzba, Study Chair — Northen state medical university
Locations (1):
- City Hospital # 1 n.a. E.E. Volosevich, Arkhangelsk, Russia

IPD SHARING:
Plan to Share IPD: No